CLINICAL TRIAL: NCT02806271
Title: Short-Term Efficacy and Mechanisms of Change of a Worry Postponement Intervention for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kathleen Tallon, Doctoral Student, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016 - 143
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: Worry Postponement; Stimulus Control
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Worry Postponement (Experimental): Two weeks of daily worry postponement
  Interventions: Behavioral: Worry Postponement; Behavioral: Worry Monitoring
- Worry Monitoring (Active Comparator): Two weeks of daily worry monitoring
  Interventions: Behavioral: Worry Monitoring
- Assessment Only Control (No Intervention): No intervention, participants will complete three assessment time points

INTERVENTIONS:
Behavioral: Worry Postponement — In worry postponement, participants are instructed to learn to notice naturally occurring episodes of worry. When they notice they are worrying they are instructed to disengage from their worry and postpone it to a designated 30 minute "worry period" to be carried out at the same time and place daily during the two week intervention. Participants are to use their worry time to worry about problems that have come up during the day and to problem solve where appropriate.
  Other Names: Stimulus Control for Worry
  Arms: Worry Postponement
Behavioral: Worry Monitoring — For two weeks participants are instructed to monitor their worry using a smartphone based application. Participants are instructed to make a record each time they have a worry episode by briefly describing the content of their worry. Participants also complete two brief daily questionnaires about the duration of their worry, the intensity of their worry, their ability to disengage from their worry, and the occurrence of nighttime episodes of worry.
  Arms: Worry Monitoring; Worry Postponement

SUMMARY:
Worry postponement is a commonly recommended treatment component in cognitive behavioral therapy for Generalized Anxiety Disorder in which people are asked to postpone naturally occurring instances of worry to a designated 30 minute "worry period" later in the day. Despite being commonly recommended, there is little known about the efficacy and mechanisms of worry postponement. The purpose of this study is to determine the efficacy and mechanisms of change of a two-week worry postponement intervention in people with Generalized Anxiety Disorder. Ninety subjects with generalized anxiety disorder will be randomly assigned to two weeks of daily worry postponement, two weeks of worry monitoring, or an assessment only control condition. Changes in worry or associated features will be examined at post intervention and at a 2-week follow up.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is a disorder characterized by excessive and uncontrollable worry. People with GAD report that worry significantly interferes with their ability to enjoy their life and function effectively in their roles. Worry postponement is a treatment technique developed by Borkovec and colleagues (1983) to reduce excessive worry. In worry postponement, people are instructed to notice naturally occurring episodes of worry and to then disengage from their worry and postpone it to a designated 30 minute "worry period" later in the day. People are instructed to confine their worry to this 30 minute period and to use that period to problem solve concerns they have been having. Worry postponement is a widely recommended technique for treating excessive worry in people with GAD and is often combined with other cognitive-behavioural interventions. Despite being commonly recommended, there are very few studies demonstrating worry postponement's efficacy for reducing worry, and no studies have looked at the effect of this intervention in people with GAD. The present study aims to extend the literature by comparing a two-week worry postponement intervention to worry monitoring alone and to an assessment only control condition. Participants will complete baseline self-report measures of worry and associated symptoms and cognitive processes. They will complete three computer tasks measuring attention control. They will then be randomized to one of three conditions (worry postponement, worry monitoring, assessment only control). Participants will follow instructions corresponding to their condition daily for two weeks. In the worry postponement and worry monitoring conditions this will involve completing brief daily worry questionnaires at home for the two weeks of the intervention. In the assessment only condition participants will not complete any measures during the two weeks after the first session. Subsequent to this, all participants will return to the lab to repeat baseline measures, and will return again two weeks later to complete measures. The entire study will require three lab visits, spanning over four weeks. This study aims to determine what the effects of worry postponement are, relative to worry monitoring and assessment only, on worry, GAD and associated symptoms, and cognitive processes related to worry. A secondary aim of this study is to examine which mechanisms predict change in worry in a worry postponement study. This will be the first study to our knowledge, to examine these questions in a sample of people with GAD. This study will provide important information for optimizing the treatment of worry in people with GAD.

ELIGIBILITY:
Inclusion Criteria:

1. Endorse symptoms consistent with a primary diagnosis of Generalized Anxiety Disorder (GAD) as defined by DSM-5 (APA, 2013), with a clinician severity rating (CSR) ≥ 4
2. If a comorbid diagnosis is present, its associated CSR is at least 1 point lower than that of their GAD diagnosis.

Exclusion Criteria:

1. Have a current or past history of psychosis or mania, or endorse symptoms consistent with a diagnosis of a substance use disorder in the past 12 months
2. Report clinically significant suicidal ideation, intent, or plan
3. Participants will be excluded if they are currently receiving psychological treatment or counseling (e.g., cognitive behaviour therapy, supportive counseling, etc.), unless this treatment is infrequent (meeting once monthly or less) or the participant has been receiving consistent weekly treatment for 12 weeks and still meets all other eligibility criteria
4. Are taking psychotropic medications and have had a change in dose in the past 12 weeks. If they have recently discontinued a psychotropic medication, they will be included if it has been at least 1 month since discontinuation, or 3 months if they had been taking fluoxetine/Prozac. If a participant is taking psychotropic medication on an as needed basis (e.g., benzodiazepines), they will be included and their use of this medication will be noted in order to assess whether it has a moderating effect on intervention outcome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in worry as measures by the Penn State Worry Questionnaire - Past Week | This measure will be administered four times over the course of the four week study; changes will be examined in scores from baseline, at 1 week (mid-intervention), at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)

SECONDARY OUTCOMES:
Change in mindfulness the Cognitive and Affective Mindfulness Scale-Revised | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in mindfulness as measured by the Southampton Mindfulness Questionnaire | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in problem solving as measured by Social Problem Solving Inventory - Revised | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in cognitive avoidance as measured by the Cognitive Avoidance Questionnaire | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in attentional control as measured by the Random Interval Generation Task | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in attentional control as measured by the N-back task | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in worry frequency as measured by daily worry diaries | Worry measures completed daily during two week intervention period
Change in meta cognitive beliefs about worry as measured by the Metacognitions Questionnaire-30 | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in attentional control over worry as measured by the Breathing Focus Task | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in symptoms of depression as measured by the Depression, Anxiety, and Stress Scales - 21 | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in symptoms of anxiety as measured by the Depression, Anxiety, and Stress Scales - 21 | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in symptoms of insomnia as measured by the Insomnia Severity Index | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in health complaints as measured by the Subjective Health Complaints Questionnaire | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)
Change in rumination as measured by the Ruminative Response Scales | This measure will be administered three times over the course of the four week study; changes will be examined in scores from baseline, at 2 weeks (immediately post intervention), and at 4 weeks (2 week follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Tallon, MA, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be disseminated via conference presentations, journal publications, and through our lab website. Upon request anonymized individual participant data may be made available to a publishing journal or individual research group. Individual research groups interested in accessing anonymized data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and CVs. Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal.

REFERENCES:
- [Background] Borkovec TD, Wilkinson L, Folensbee R, Lerman C. Stimulus control applications to the treatment of worry. Behav Res Ther. 1983;21(3):247-51. doi: 10.1016/0005-7967(83)90206-1. No abstract available. PMID 6615390
- [Background] Brosschot JF, Van Der Doef M. Daily worrying and somatic health complaints: Testing the effectiveness of a simple worry reduction intervention. Psychol Health. 2006; 21: 19-31. doi:10.1080/14768320500105346
- [Background] McGowan SK, Behar E. A preliminary investigation of stimulus control training for worry: effects on anxiety and insomnia. Behav Modif. 2013 Jan;37(1):90-112. doi: 10.1177/0145445512455661. Epub 2012 Sep 12. PMID 22977265
- [Background] Newman MG, Borkovec TD. Cognitive behavioral therapy for worry and generalized anxiety disorder. In: Simos G, editor. Cognitive behaviour therapy: A guide for the practising clinician. New York; Taylor & Francis; 2002. P 150-172.
- See also: Lab website — http://psychlabs.ryerson.ca/caplab/